CLINICAL TRIAL: NCT01233544
Title: The International Liver Tumor Group RAS-trial Radiofrequency Ablation Versus Stereotactic Body Radiation Therapy for Colorectal Liver Metastases: A Randomized Trial
Brief Title: Radiofrequency Ablation Versus Stereotactic Radiotherapy in Colorectal Liver Metastases
Acronym: RAS01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: University of Aarhus (Other)
Collaborators: Danish Center for Interventional Research in Radiation Oncology (CIRRO) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAS 01
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Carcinoma; Liver Metastases
Keywords: Colorectal carcinoma; Liver metastases; Stereotactic body radiation therapy; Radiofrequency ablation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stereotactic body radiation therapy (Experimental): Colorectal liver metastases treated by SBRT
  Interventions: Procedure: SBRT or RFA
- Radiofrequency ablation (Active Comparator): Colorectal liver metastases treated by RFA
  Interventions: Procedure: SBRT or RFA

INTERVENTIONS:
Procedure: SBRT or RFA — Patients are allocated to one of the two arms in a 1:1 randomization
  Other Names: Stereotactic body radiation therapy; Radiofrequency ablation

SUMMARY:
This randomized clinical phase III trial is testing the efficacy of radiofrequency ablation (RFA) and stereotactic body radiotherapy (SBRT) in the treatment of colorectal carcinoma liver metastases.

Primary end point is local progression free survival.

DETAILED DESCRIPTION:
Patients with 1-4 inoperable colorectal liver metastases, no more 4 cm in diameter are randomized to either RFA or SBRT. Primary end point i local progression free survival. Chemotherapy is allowed before and after study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the colon or rectum
* Liver metastases
* Inoperable (technical or medical)
* 1-4 metastases
* Maximum 40 mm in diameter
* Suitable for both therapies, RFA and SBRT

Exclusion Criteria:

* Uncontrolled extrahepatic disease and uncontrolled primary cancer
* Liver cirrhosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Local progression-free survival | 3 years

SECONDARY OUTCOMES:
Toxicity | 3 years
Survival | 3 years
Progression (local or distant) | 3 years
Quality of life | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Morten Høyer, MD PhD, Principal Investigator — Aarhus University Hospital
Locations (2):
- Aarhus University Hospital, Aarhus C, Denmark
- Karolinska Institute, Huddinge, Stockholm, Sweden

REFERENCES:
- See also: Centre for Interventional Research in Radiation Oncology — http://www.cirro.dk